CLINICAL TRIAL: NCT05273658
Title: Effects of Cannabis/Alcohol on Driving Performance and Field Sobriety Tests
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Termination of funding
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Thomas D. Marcotte, PhD, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 192048
Record Dates: First submitted 2022-02-28; First posted 2022-03-10 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Driving Impaired; Alcohol Intoxication; Driving Under the Influence; Cannabis Intoxication
Keywords: Cannabis; Alcohol; Driving
MeSH Terms: conditions — Alcoholic Intoxication; Driving Under the Influence; Marijuana Abuse | interventions — nabiximols; Ethanol

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to smoke a cannabis cigarette containing placebo (.02%) or 18.1% THC, and consume alcohol to achieve a breath alcohol level of .07, .10, or 0.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Cannabis will be dispensed from the Research Pharmacy. Alcohol will be dispensed by a research staff member who is not involved in any assessments. All assessors, investigators, and participants are blinded to the THC and alcohol content.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo cannabis and placebo alcohol
  Interventions: Drug: Cannabis; Drug: Alcohol
- Cannabis, No alcohol (Experimental): 18.16% THC, placebo alcohol
  Interventions: Drug: Cannabis; Drug: Alcohol
- Cannabis, Low dose alcohol (Experimental): 18.16% THC, .07 breath alcohol concentration
  Interventions: Drug: Cannabis; Drug: Alcohol
- Placebo cannabis, High dose alcohol (Experimental): <.1% THC, .10 Breath alcohol concentration
  Interventions: Drug: Cannabis; Drug: Alcohol
- Placebo cannabis, Low dose alcohol (Experimental): <.1% THC, .07 breath alcohol concentration
  Interventions: Drug: Cannabis; Drug: Alcohol

INTERVENTIONS:
Drug: Cannabis — Participants will smoke a cannabis cigarette ad libitum as per their usual routine
  Other Names: Marijuana
Drug: Alcohol — Participants will ingest alcohol to achieve the target breath alcohol level

SUMMARY:
The overarching aim of this study is to examine the impact of acute cannabis and alcohol administration on driving performance, as well as identify methods for detecting driving under the influence of these substances. One-hundred twenty-five healthy volunteers will be randomized into one of 5 conditions; those who receive 1) low dose alcohol and placebo cannabis, 2) low dose alcohol and tetrahydrocannabinol (THC), 3) high dose alcohol and placebo cannabis, 4) placebo alcohol and THC, and 5) double placebo. Cannabis inhaled ad libitum and/or ingested alcohol will take place at the beginning of the day followed by the completion of driving simulations, components of the Drug Recognition Expert (DRE) evaluations, and bodily fluid draws (e.g., blood, oral fluid/saliva, breath) over the subsequent 4 hours after ingestion. The purpose of this study is to determine (1) the impact of Δ9-THC on driving performance with and without concurrent alcohol ingestion (2) the duration of driving impairment in terms of hours from initial use, (3) the relationship between performance on the DRE measures and cannabis/alcohol ingestion, and 4) if saliva or expired air can serve as a useful adjunct to the field for blood sampling.

DETAILED DESCRIPTION:
Driving under the influence of alcohol and cannabis presents significant safety risks. In the real world, impairment is usually determined via the standardized field sobriety tests (SFSTs), a series of psychophysiological tests conducted by law enforcement officers. These include the Horizontal Gaze Nystagmus (HGN; eye movements when following the officer's fingers in space), Walk and Turn (WAT; walking nine steps, turning, and walking back), and One Leg Stand (OLS; holding each leg in the air for a designated period of time).

Despite a vast literature documenting impaired driving behavior due to alcohol consumption, much less is known regarding driving under the influence of cannabis, and even less about how the combination of alcohol and cannabis may affect driving behavior. This study will examine whether either, or both, conditions significantly impact performance in a driving simulator, on cognitive measures, and during the comprehensive Drug Recognition Expert evaluations (which includes SFSTs, as well as additional measures).

Alcohol studies. Higher blood alcohol levels (BACs) have been consistently related to impaired driving. BACs greater than .08% have been associated with 5.5 times higher crash risk compared to those without alcohol or drugs. In terms of detecting alcohol-related impairment, SFSTs have consistently been shown to be predictors of a blood alcohol concentration of .08%.

Cannabis studies. Several studies suggest higher doses of whole-blood or plasma delta-9 tetrahydrocannabinol (THC) concentration are associated with increased crash risk and crash culpability. However, attempts to define a cut-off point for blood THC levels have proven to be challenging. Unlike alcohol, for which a level can be reasonably measured using a breathalyzer (and confirmed with a blood test), detection of a cut-off point for intoxication related to THC concentration has eluded scientific verification. Most recently, we did not find any correlation between blood THC concentrations and driving performance. To date, the relationship between SFSTs and cannabis use/impairment have been mixed across studies.

Cannabis and Alcohol. There have been a limited number of studies examining the combination of cannabis and alcohol on driving and/or field sobriety test performance.

With respect to subjective effects, alcohol has been found to potentiate the duration of the cannabis effects, with subjective effects being longer in the cannabis-alcohol combinations compared to either drug alone. Participants also reported more effects after alcohol and cannabis were combined, compared to alcohol alone. Another study found that alcohol pre-treatment decreased the latency to the cannabis effects, and increased the duration of the effects. It has also been hypothesized that frequent cannabis users may develop cross-tolerance to the effects of alcohol.

Some studies have found SFSTs to be only mildly sensitive to cannabis effects in heavy cannabis users, but sensitive to doses of alcohol.

There have also been suggestions that the concurrent presence of cannabis and alcohol may result in increased THC and 11-Hydroxy-Δ9-tetrahydrocannabinol (11-OH-THC) levels, possibly by affecting initial absorption (resulting in higher concentrations immediately post-inhalation; the overall area under the curve (AUC) does not differ based upon alcohol ingestion), although the possible mechanisms for this - such as increased cardiac output facilitating absorption via increased pulmonary capillary flow, or less cannabis self-titration after alcohol intake - are as yet unresolved.

Research Design

One-hundred twenty-five healthy volunteers will be randomized into one of 5 conditions; those who receive 1) low dose alcohol and placebo cannabis, 2) low dose alcohol and THC, 3) high dose alcohol and placebo cannabis, 4) placebo alcohol and THC, and 5) double placebo.

Cannabis, acquired from the National Institute on Drug Abuse Drug Supply Program, will be inhaled ad libitum and/or ingested alcohol will take place at the beginning of the day followed by the completion of driving simulations, components of the Drug Recognition Expert (DRE) evaluations, and bodily fluid draws (e.g., blood, oral fluid [OF] saliva, breath) over the subsequent 4 hours after ingestion.

Driving simulations will be conducted using a 3-monitor, fully-interactive STISIM (Systems Technology Inc. Simulator) console system. The simulations will be similar to those used in our recently completed study of 191 cannabis users.

Drug Recognition Expert (DRE) evaluations will be conducted by DREs, and will consist of 1) Preliminary Examination and First Pulse; 2) Eye Examinations: Horizontal gaze nystagmus (HGN); Vertical gaze nystagmus (VGN); Lack of convergence (LOC); 3) Divided Attention Psychophysical Tests: Modified Romberg balance; Walk and turn; One leg stand; Finger to nose; 4) Vital Signs and Second Pulse (Blood pressure, temperature, pulse); 5) Dark Room Examinations (pupillometer): Assess for dilation or constriction; pupillary response to light; 6) Examination for Muscle Tone; 7) Third Pulse.

Cannabinoids levels in blood, oral fluid, and breath will be determined via liquid chromatography with tandem mass spectrometry (LC-MS-MS).

The results of this study will further advance the understanding of the impact of acute cannabis and alcohol administration on driving performance, as well as the best methods for detecting driving under the influence of these substances.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 to 55
* Must be a licensed driver and driven a minimum of 1,000 miles in the past year
* Experience with cannabis and alcohol

Exclusion Criteria:

* At the discretion of the examining physician, individuals with significant cardiovascular, hepatic or renal disease, uncontrolled hypertension, and chronic pulmonary disease (eg, asthma, COPD) will be excluded.
* Unwillingness to abstain from cannabis for 2 days prior to screening and experimental visits
* Positive pregnancy test
* A positive result on toxicity screening for cocaine, amphetamines, opiates, and phencyclidine (PCP) will exclude individuals from participation.
* Unwilling to refrain from driving or operating heavy machinery after consuming study medication.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Composite Drive Score | Participants are assessed pre-smoking/drinking, and then approximately 30 minutes, 1 hour 30 minutes, and 3 hours 30 minutes post-smoking
  The Composite Drive Score (CDS) is a z-score comprised of key variables from the simulator tasks (SDLP, speed deviation, and task accuracy during the modified Surrogate Reference Task (mSuRT); coherence from the car following task). This outcome reflects the change in CDS from the pre-smoking assessment, at each timepoint.
  The z-score indicates the number of standard deviations away from the mean from the baseline performance for the entire group. A Z-score of 0 is equal to the mean of a reference population (in this case the pre-smoking performance for the entire group).
  Higher z-scores at each timepoint indicate worse performance (variables that went in the opposite direction were reflected in order to have all variables have the same direction). When examining the change in Composite Drive Score (this outcome variable), a higher score indicates a decline in performance (e.g., Time 2 minus Time1).

SECONDARY OUTCOMES:
DRE Impairment | Approximately 1.5 hours and 2.5 hours after alcohol/cannabis administration
  DRE officers' determination regarding participant impairment
Whole blood THC concentration | Approximately 30 minutes after alcohol/cannabis administration
  Whole blood THC concentrations determine via LC-MS-MS
Oral Fluid THC concentration | Approximately 30 minutes after alcohol/cannabis administration
  Oral fluid THC concentrations determine via LC-MS-MS
Breath THC concentration | Approximately 30 minutes after alcohol/cannabis administration
  Breath THC concentrations determine via LC-MS-MS

REFERENCES:
- [Result] Movig KL, Mathijssen MP, Nagel PH, van Egmond T, de Gier JJ, Leufkens HG, Egberts AC. Psychoactive substance use and the risk of motor vehicle accidents. Accid Anal Prev. 2004 Jul;36(4):631-6. doi: 10.1016/S0001-4575(03)00084-8. PMID 15094417
- [Result] Stuster J. Validation of the standardized field sobriety test battery at 0.08% blood alcohol concentration. Hum Factors. 2006 Fall;48(3):608-14. doi: 10.1518/001872006778606895. PMID 17063973
- [Result] Grotenhermen F, Leson G, Berghaus G, Drummer OH, Kruger HP, Longo M, Moskowitz H, Perrine B, Ramaekers JG, Smiley A, Tunbridge R. Developing limits for driving under cannabis. Addiction. 2007 Dec;102(12):1910-7. doi: 10.1111/j.1360-0443.2007.02009.x. Epub 2007 Oct 4. PMID 17916224
- [Result] Hartman RL, Brown TL, Milavetz G, Spurgin A, Gorelick DA, Gaffney G, Huestis MA. Controlled vaporized cannabis, with and without alcohol: subjective effects and oral fluid-blood cannabinoid relationships. Drug Test Anal. 2016 Jul;8(7):690-701. doi: 10.1002/dta.1839. Epub 2015 Aug 10. PMID 26257143
- [Result] Ramaekers JG, Theunissen EL, de Brouwer M, Toennes SW, Moeller MR, Kauert G. Tolerance and cross-tolerance to neurocognitive effects of THC and alcohol in heavy cannabis users. Psychopharmacology (Berl). 2011 Mar;214(2):391-401. doi: 10.1007/s00213-010-2042-1. Epub 2010 Oct 30. PMID 21049267
- [Result] Hartman RL, Brown TL, Milavetz G, Spurgin A, Pierce RS, Gorelick DA, Gaffney G, Huestis MA. Cannabis effects on driving lateral control with and without alcohol. Drug Alcohol Depend. 2015 Sep 1;154:25-37. doi: 10.1016/j.drugalcdep.2015.06.015. Epub 2015 Jun 23. PMID 26144593
- [Result] Hoffman MA, Hubbard JA, Sobolesky PM, Smith BE, Suhandynata RT, Sanford S, Sones EG, Ellis S, Umlauf A, Huestis MA, Grelotti DJ, Grant I, Marcotte TD, Fitzgerald RL. Blood and Oral Fluid Cannabinoid Profiles of Frequent and Occasional Cannabis Smokers. J Anal Toxicol. 2021 Sep 17;45(8):851-862. doi: 10.1093/jat/bkab078. PMID 34173005
- [Result] Hubbard JA, Smith BE, Sobolesky PM, Kim S, Hoffman MA, Stone J, Huestis MA, Grelotti DJ, Grant I, Marcotte TD, Fitzgerald RL. Validation of a liquid chromatography tandem mass spectrometry (LC-MS/MS) method to detect cannabinoids in whole blood and breath. Clin Chem Lab Med. 2020 Apr 28;58(5):673-681. doi: 10.1515/cclm-2019-0600. PMID 31527291